CLINICAL TRIAL: NCT06293924
Title: The Pericardial Fluid Analysis in Recurrent Pericarditis Trial
Brief Title: Pericardial Fluid Analysis in Recurrent Pericarditis
Acronym: PEFLANA
Status: Enrolling by invitation | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Enrico Tombetti, Co-Principal Investigator, ASST Fatebenefratelli Sacco
Other Study IDs: The PEFLANA Trial
Record Dates: First submitted 2024-02-26; First posted 2024-03-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Acute Pericarditis; Pericardial Effusion; Pericardial Disease; Pericardial Fluid Exudate; Autoinflammatory Disorders; Autoinflammatory Disease
Keywords: Acute Pericarditis; Recurrent Pericarditis; Pericardial Effusion; Pericardiocentesis; Cardiac surgery; Cytofluorometry; Gene expression analysis; Autoinflammatory Disorders
MeSH Terms: conditions — Pericardial Effusion; Pericarditis | interventions — Pericardiocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Pericarditis patients: Patients with acute idiopathic or post-cardiac injury pericarditis who require diagnostic or therapeutic pericardiocentesis. Four ml of pericardial fluid should be collected: 2 ml for biochemical analysis in lithium heparin or serum-gel separator-associated tubes, and 2 ml for cellular analysis in K3 ethylenediaminetetraacetic acid (K3-EDTA) tubes.
  Interventions: Diagnostic Test: Pericardiocentesis; Diagnostic Test: Cytofluorometry and Gene expression analysis
- Pericardial effusion patients without inflammation: Subjects with non-inflammatory pericardial effusion who require diagnostic or therapeutic pericardiocentesis. Four ml of pericardial fluid should be collected: 2 ml for biochemical analysis in lithium heparin or serum-gel separator-associated tubes, and 2 ml for cellular analysis in K3 EDTA tubes.
  Interventions: Diagnostic Test: Pericardiocentesis; Diagnostic Test: Cytofluorometry and Gene expression analysis
- Cardiac surgery pericardial effusion: Patients who undergo cardiac surgery that involves a pericardiotomy. During cardiac surgery, 4 ml of pericardial fluid is collected and analyzed upon opening the pericardial sac. Four ml of pericardial fluid should be collected: 2 ml for biochemical analysis in lithium heparin or serum-gel separator-associated tubes, and 2 ml for cellular analysis in K3 EDTA tubes.
  Interventions: Diagnostic Test: Pericardiotomy; Diagnostic Test: Cytofluorometry and Gene expression analysis

INTERVENTIONS:
Diagnostic Test: Pericardiocentesis — Enrolled patients will not undergo any invasive investigations outside of normal clinical practice. Patients with acute pericarditis and non-inflammatory pericardial effusion will undergo pericardiocentesis for diagnostic or therapeutic purposes.
  Four ml of pericardial fluid will be collected: 2 ml for biochemical analysis in lithium heparin or serum-gel separator-associated tubes, and 2 ml for cellular analysis in K3 EDTA tubes.
  Groups: Pericardial effusion patients without inflammation; Pericarditis patients
Diagnostic Test: Pericardiotomy — During any type of cardiac surgery involving pericardiotomy, 4 ml of pericardial fluid will be collected and analyzed upon opening the pericardial sac of enrolled patients.
  Four ml of pericardial fluid will be collected: 2 ml for biochemical analysis in lithium heparin or serum-gel separator-associated tubes, and 2 ml for cellular analysis in K3 EDTA tubes.
  Groups: Cardiac surgery pericardial effusion
Diagnostic Test: Cytofluorometry and Gene expression analysis — A 30 ml sample of peripheral venous blood in K3 EDTA tubes will be collected by enrolled patients who participating in the translational substudy and stored with pericardial fluid samples.
  Pericardial fluid cells by lineage and expression of inflammatory cytokines will be characterized through cytofluorometry and expression profile analysis of transcribed RNAs. Cytokine concentrations in peripheral blood and pericardial fluid will be analyzed by molecular assay. Peripheral blood mononucleated cells (PBMCs) and pericardial fluid cells will be cultured in vitro and exposed to the main therapies used during pericarditis, to verify the effects on gene expression and inflammatory molecules.

SUMMARY:
This clinical trial aims to examine the biochemical and cytological features of pericardial effusion during acute and recurrent pericarditis and to understand the molecular factors responsible for pathogenesis. The primary objective of this study is to identify and validate diagnostic criteria in pericardial fluid analysis that can differentiate patients with acute and recurrent pericarditis from those with only pericardial fluid but no inflammation.

This study will enroll patients with acute pericarditis who require pericardiocentesis for either diagnostic or therapeutic purposes. Two control groups will also be included: one consisting of patients who need cardiac surgery with a collection of pericardial fluid, and the other consisting of patients who require pericardiocentesis for non-inflammatory pericardial effusion. The purpose of the study is to compare the cell activation status and cytokines present in pericardial fluid during acute pericarditis with those present during other pericardial pathologies.

DETAILED DESCRIPTION:
Idiopathic recurrent pericarditis is a condition characterized by recurrent inflammation of the pericardial sac and sometimes another serosa, accompanied by systemic signs and symptoms. Differential diagnosis of this condition includes all forms of pericarditis secondary to other diseases such as infections, autoimmune and autoinflammatory diseases, malignancy and other conditions (post-actinic, post-traumatic, post-pericardiotomy or post-infarct pericarditis, or those associated with metabolic dysregulations such as uremia). Some patients have pericardial effusion without any signs of inflammation: this condition is known as idiopathic pericardial effusion.

The analysis of pericardial effusion helps diagnostic and therapeutic decisions. European Society of Cardiology (ESC) guidelines recommend pericardial fluid analysis from pericardiocentesis or surgical access only whenever a suspected infectious or neoplastic form. Pericardiocentesis is also a procedure used to remove excess fluid from the sac surrounding the heart with hemodynamic effects on ventricular diastolic filling. It is performed in emergencies such as cardiac tamponade to relieve pressure on the heart.

The causes and mechanisms of idiopathic pericarditis are not yet well understood. However, studies have shown that colchicine, a medication used to treat this condition, can prevent the formation of microtubules, the migration of neutrophils, and the formation of the NLRP3 inflammasome. These factors have been suggested to play a role in the development of this disease. In addition, research has focused on the use of Anakinra, an anti-interleukin 1 (IL-1) drug, in the treatment of acute pericarditis. This confirms the possible involvement of IL-1 beta in this disease. It is produced by the activation of a complex called NLRP3 inflammasome, which is triggered by microbial products (PAMPs), urate crystals, cholesterol, and molecules known as damage-associated molecular patterns (DAMPs). Therapeutic options for idiopathic pericarditis include colchicine, non-steroidal anti-inflammatory drugs (NSAIDs), steroids, and IL-1 antagonists to regulate inflammation and leukocyte migration.

This study focuses on two main unmet needs related to acute and recurrent pericarditis. The first need is related to the informativeness of the data obtained through pericardiocentesis. Although the biochemical analysis is recommended by ESC guidelines, the most valuable data in the diagnostic process comes from cytological and microbiological analyses. These analyses help in excluding neoplastic or infectious etiologies. Biochemical features of pericardial fluid are less understood than those of peritoneal and pleural fluids. Specific biochemical parameters used to distinguish exudation as Light's criteria do not apply to pericardial fluid: a previous study showed a unique composition of pericardial fluid, which suggests that Light's criteria cannot be used in this case. The second unsatisfied need is related to pathogenesis, including the pathway of Interleukin-1 (IL-1) at the level of pericardial fluid and which cells are responsible for local cytokines and inflammatory mediators productions.

This study aims to collect observational data on pericardial effusion analysis and to analyse cellular and molecular composition in a subgroup of patients to assess the pathophysiological mechanisms of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute idiopathic or post-cardiac injury pericarditis who require diagnostic or therapeutic pericardiocentesis (Interventional arm)
* Subjects with non-inflammatory pericardial effusion who require diagnostic or therapeutic pericardiocentesis (First control arm)
* Patients who undergo cardiac surgery that involves a pericardiotomy (Second control arm)

Exclusion Criteria:

* Pregnancy or breastfeeding
* Ongoing infections, including active viral hepatitis or Coronavirus Disease 19 (COVID-19) positivity in the previous 21 days
* Systemic inflammatory disorders not attributable to pericarditis, excluding inflammatory diseases in remission
* Solid or haematological malignancies, ongoing or less than 6 months disease-free interval or anti-blastic chemotherapy (excluding the hormone therapy)
* Immunosuppressive therapy for reasons other than pericarditis treatment.
* Moderate-severe kidney failure (GFR < 30 ml/min)
* Moderate-severe liver failure (Child-Pug B or C), active hepatitis
* Diabetes mellitus
* Severe hypoproteinemia/malnutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the first two arms, patients from the primary care clinic (Emergency room department). For the third arm, patients who need to undergo cardiac surgery with pericardial sac involvement.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Differences in cell counts among inflammatory and non-inflammatory pericardial effusion. | 48 months from patient's enrollment
  Both automated cytometry and manual counting were used to obtain absolute and relative cell counts from peripheral blood samples and pericardial fluids. It can help identify and establish diagnostic criteria for distinguishing between patients with acute or recurrent pericarditis and those with non-inflammatory pericardial fluid.
Difference in biochemical parameters among inflammatory and non-inflammatory pericardial effusion | 48 months from patient's enrollment
  This analysis evaluates the differences in pericardial fluid and peripheral blood among biochemical parameters (total proteins and albumin, lactate dehydrogenase, blood glucose, and cholesterol concentrations). It can help distinguish between patients with acute or recurrent pericarditis and those with non-inflammatory pericardial fluid, thereby aiding in the validation of diagnostic criteria.

SECONDARY OUTCOMES:
Difference of IL-1 expression in pericardial fluid cells among inflammatory and non-inflammatory pericardial effusion | 48 months from patient's enrollment
  A flow cytometry analysis is performed to assess absolute and relative cell counts expressing IL-1 in pericardial fluid for the differentiation between pericarditis and non-inflammatory pericardial fluid.
Differences of inflammatory cytokine expression in pericardial fluid cells among inflammatory and non-inflammatory pericardial effusion | 48 months from patient's enrollment
  A flow cytometry analysis is performed to assess absolute and relative cell counts expressing inflammatory cytokines in pericardial fluid for the differentiation between pericarditis and non-inflammatory pericardial fluid.
Differences of gene expression in pericardial fluid cells among inflammatory and non-inflammatory pericardial effusion | 48 months from patient's enrollment
  A gene expression analysis using transcribed RNA assesses absolute and relative cell counts expressing inflammatory cytokines in pericardial fluid and blood samples for the differentiation between pericarditis and non-inflammatory pericardial fluid.
Differences of gene expression in pericardial fluid and blood cells during pericarditis | 48 months from patient's enrollment
  A gene expression analysis evaluates the increase of activated inflammatory cells in pericarditis through absolute and relative cell counts in pericardial fluid and blood samples using transcribed RNA. This analysis can confirm the correlation between activated inflammatory cells in pericardial and blood samples during pericarditis.
Differences in cytokine and other molecule concentrations between pericardial fluid and blood cells in pericarditis | 48 months from patient's enrollment
  Biochemical analysis evaluates the increase of inflammatory cytokines and other molecules in pericarditis in pericardial fluid and blood samples using normal methods of analysis. This analysis can confirm the correlation between inflammatory mediators in pericardial and blood samples during pericarditis.
Correlation of inflammatory mediators in pericardial fluid and clinical features during pericarditis | 48 months from patient's enrollment
  Biochemical analysis evaluates the increase of inflammatory cytokines and other molecules in pericarditis in pericardial fluid and blood samples. This analysis can confirm the correlation between cytokines and other molecules and clinical manifestations during pericarditis.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Luca Brucato, Prof., Principal Investigator — ASST Fatebenefratelli Sacco
Locations (1):
- ASST FAtebenefratelli Sacco, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No